CLINICAL TRIAL: NCT07374614
Title: An Observational Study of the Efficacy and Safety of Iruplinalkib(WX-0593) in ALK-positive Advanced Lung Adenocarcinoma Following Lorlatinib Treatment
Brief Title: Iruplinalkib in ALK-Positive Advanced Lung Adenocarcinoma After Lorlatinib
Acronym: SAILOR
Status: Recruiting | Type: Observational
Sponsor: Peking University Shenzhen Hospital (Other)
Collaborators: Shenzhen People's Hospital (Other); Longgang District People's Hospital of Shenzhen (Other); Sun Yat-sen University Cancer Hosptial (Unknown); Eighth Affiliated Hospital, Sun Yat-sen University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); People Hospital of New District Longhua Shenzhen (Unknown)
Responsible Party: Principal Investigator, Fen Wang, Associate chief physician, Peking University Shenzhen Hospital
Other Study IDs: 2025-324
Record Dates: First submitted 2026-01-16; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer; ALK; Iruplinalkib; Lorlatinib; Real-world Study; Observational Study
Keywords: Iruplinalkib; ALK-postive; Post-Lorlatinib; Advanced Lung Adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Treatment group
  Interventions: Drug: Iruplinalkib tablets

INTERVENTIONS:
Drug: Iruplinalkib tablets — 180mg, QD

SUMMARY:
This observational study aims to evaluate the real-world effectiveness and safety of iruplinalkib in patients with advanced ALK-positive lung adenocarcinoma who have progressed on or are intolerant to prior lorlatinib therapy. The results are expected to provide real-world evidence to inform clinical decision-making for this heavily pretreated patient population.

DETAILED DESCRIPTION:
Background & Unmet Need:

Lorlatinib, a third-generation ALK tyrosine kinase inhibitor (TKI), is a standard treatment option for patients with advanced ALK-positive lung adenocarcinoma, particularly following the failure of earlier-generation ALK inhibitors. Despite its potent central nervous system penetration and broad coverage of ALK resistance mutations, acquired resistance and disease progression remain inevitable for most patients. Currently, there is no established standard of care for patients who progress on lorlatinib, representing a significant unmet clinical need.

Rationale for Iruplinalkib:

Iruplinalkib is a novel ALK inhibitor exhibiting high selectivity and activity against a broad spectrum of ALK resistance mutations, including those associated with resistance to prior ALK TKIs. While preliminary clinical studies have demonstrated promising antitumor activity and a manageable safety profile in patients with ALK-positive non-small cell lung cancer (NSCLC), data specifically evaluating iruplinalkib in the post-lorlatinib setting are limited, particularly within real-world clinical practice.

Study Objectives:

This study is designed as an observational investigation to assess the real-world effectiveness and safety of iruplinalkib in patients with advanced ALK-positive lung adenocarcinoma who have received prior lorlatinib treatment. The study will include eligible patients who are prescribed iruplinalkib as part of routine clinical practice. This study aims to characterize the clinical benefit of iruplinalkib and explore its potential role as a subsequent-line treatment option in this specific population.

ELIGIBILITY:
Inclusion Criteria:

1. Population: Male or female patients aged ≥18 years.
2. Diagnosis: Histologically or cytologically confirmed advanced lung adenocarcinoma.
3. Molecular Status: Documentation of ALK rearrangement confirmed by a validated test (e.g., NGS, IHC, FISH).
4. Prior Therapy: Prior treatment with lorlatinib (in any line of therapy), with documented disease progression or intolerance.
5. Current Therapy: Initiated treatment with iruplinalkib in the real-world setting.
6. Measurability: Presence of at least one evaluable lesion (measurable or non-measurable) for response assessment.
7. Data Availability: availability of key clinical data (baseline characteristics, treatment history, and follow-up outcomes).

Exclusion Criteria:

1. Lack of Exposure: Patients who never actually received iruplinalkib or took only a trivial amount (e.g., < 1 week/cycle) before withdrawal for non-medical reasons.
2. Wrong Diagnosis: Active malignancy of other histological types (excluding treated basal cell carcinoma, etc.).
3. Confounding: Participation in another interventional clinical trial involving an investigational anti-tumor drug concurrently.
4. Pregnancy: Pregnant or breastfeeding women.
5. Data Quality: Missing critical medical records that preclude assessment of primary endpoints (e.g., unknown start date, unknown prior therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALK-positive lung adenocarcinoma patients who receive Iruplinalkib after lorlatinib treatment.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Real-World Progression-Free Survival (rwPFS) | From index date through study completion, an average of 36 months
  Time from treatment initiation to the earliest of death or clinical disease progression. Progression is defined by the treating provider's assessment recorded in the medical record, based on radiology, laboratory, or physical exam findings, distinct from RECIST-based radiographic progression.

SECONDARY OUTCOMES:
Time to Next Treatment (TTNT) | From index date to the start of next line of therapy, assessed up to 36 months
  TTNT is defined as the time interval from the index date (date of first dose of the study treatment) to the date of the first administration of a new (subsequent) systemic anti-cancer therapy. This outcome distinguishes the duration of the current line of therapy before a switch is made. Patients who die without receiving a subsequent therapy are censored at the date of death. Patients who remain on the study treatment or discontinue treatment without starting a new line are censored at their last known activity date or the data cutoff date.
Overall survival (OS) | From index date through study completion, an average of 36 months
  To assess overall survival, define as first dose to the death of the subject due to any cause
Treatment-related adverse reactions ( TRAE ) | From the index date through the date of Iruplinalkib discontinuation or the start of a new anti-cancer therapy (whichever occurs first), assessed up to 36 months.
  All AEs will be evaluated by the investigators to determine their potential relationship to iruplinalkib treatment based on clinical judgment, temporal association, and alternative etiologies. Events assessed as possibly, probably, or definitely related to iruplinalkib will be classified as treatment-related adverse reactions (TRAEs). The TRAEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE, 5.0). Serious adverse events (SAEs) will be identified and recorded in accordance with standard definitions or are considered medically significant by the investigator.

OTHER OUTCOMES:
Real-World Objective Response Rate (rwORR) | From index date until disease progression or start of new anti-cancer therapy, assessed up to 36 months
  rwORR is defined as the proportion of patients with a best overall response (BOR) of real-world complete response (rwCR) or real-world partial response (rwPR) as documented in the electronic health records (EHR). Response assessment is based on the treating clinician's qualitative assessment in clinical notes (clinician-anchored) and/or radiology reports, without strictly requiring RECIST 1.1 measurements. Patients without sufficient data to assess response are considered non-responders.
Real-World Disease Control Rate (rwDCR) | from index date until disease progression or start of new anti-cancer therapy, assessed up to 36 months
  rwDCR is defined as the proportion of patients with a best overall response (BOR) of real-world complete response (rwCR), real-world partial response (rwPR), or real-world stable disease (rwSD). To be classified as rwSD, the condition must be maintained for a minimum duration (e.g., at least 6 weeks) from the index date. Assessment is derived from unstructured clinical notes (clinician-anchored).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Shenzhen Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shi Y, Fang J, Hao X, Zhang S, Liu Y, Wang L, Chen J, Hu Y, Hang X, Li J, Liu C, Zhang Y, Wang Z, Hu Y, Gu K, Huang J, Zhang L, Shan J, Ouyang W, Zhao Y, Zhuang W, Yu Y, Zhao J, Zhang H, Lu P, Li W, Si M, Ge M, Geng H. Safety and activity of WX-0593 (Iruplinalkib) in patients with ALK- or ROS1-rearranged advanced non-small cell lung cancer: a phase 1 dose-escalation and dose-expansion trial. Signal Transduct Target Ther. 2022 Jan 28;7(1):25. doi: 10.1038/s41392-021-00841-8. PMID 35087031
- [Result] Camidge DR, Kim HR, Ahn MJ, Yang JCH, Han JY, Hochmair MJ, Lee KH, Delmonte A, Garcia Campelo MR, Kim DW, Griesinger F, Felip E, Califano R, Spira A, Gettinger SN, Tiseo M, Lin HM, Gupta N, Hanley MJ, Ni Q, Zhang P, Popat S. Brigatinib Versus Crizotinib in Advanced ALK Inhibitor-Naive ALK-Positive Non-Small Cell Lung Cancer: Second Interim Analysis of the Phase III ALTA-1L Trial. J Clin Oncol. 2020 Nov 1;38(31):3592-3603. doi: 10.1200/JCO.20.00505. Epub 2020 Aug 11. PMID 32780660
- [Result] Mok T, Camidge DR, Gadgeel SM, Rosell R, Dziadziuszko R, Kim DW, Perol M, Ou SI, Ahn JS, Shaw AT, Bordogna W, Smoljanovic V, Hilton M, Ruf T, Noe J, Peters S. Updated overall survival and final progression-free survival data for patients with treatment-naive advanced ALK-positive non-small-cell lung cancer in the ALEX study. Ann Oncol. 2020 Aug;31(8):1056-1064. doi: 10.1016/j.annonc.2020.04.478. Epub 2020 May 11. PMID 32418886
- [Result] Zhang S, Anjum R, Squillace R, Nadworny S, Zhou T, Keats J, Ning Y, Wardwell SD, Miller D, Song Y, Eichinger L, Moran L, Huang WS, Liu S, Zou D, Wang Y, Mohemmad Q, Jang HG, Ye E, Narasimhan N, Wang F, Miret J, Zhu X, Clackson T, Dalgarno D, Shakespeare WC, Rivera VM. The Potent ALK Inhibitor Brigatinib (AP26113) Overcomes Mechanisms of Resistance to First- and Second-Generation ALK Inhibitors in Preclinical Models. Clin Cancer Res. 2016 Nov 15;22(22):5527-5538. doi: 10.1158/1078-0432.CCR-16-0569. Epub 2016 Oct 25. PMID 27780853
- [Result] Solomon BJ, Mok T, Kim DW, Wu YL, Nakagawa K, Mekhail T, Felip E, Cappuzzo F, Paolini J, Usari T, Iyer S, Reisman A, Wilner KD, Tursi J, Blackhall F; PROFILE 1014 Investigators. First-line crizotinib versus chemotherapy in ALK-positive lung cancer. N Engl J Med. 2014 Dec 4;371(23):2167-77. doi: 10.1056/NEJMoa1408440. PMID 25470694
- [Result] Raskova Kafkova L, Mierzwicka JM, Chakraborty P, Jakubec P, Fischer O, Skarda J, Maly P, Raska M. NSCLC: from tumorigenesis, immune checkpoint misuse to current and future targeted therapy. Front Immunol. 2024 Feb 7;15:1342086. doi: 10.3389/fimmu.2024.1342086. eCollection 2024. PMID 38384472
- [Result] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751